CLINICAL TRIAL: NCT00769197
Title: Optic Nerve Head Morphology in Children With Perinatal Onset Static Encephalopathy
Brief Title: Optic Discs in Children With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Deepta Ghate MD, University of Mississippi Medical Center
Other Study IDs: 2008-0082
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2009-04-29 (Estimated); Status verified 2009-04

CONDITIONS: Cerebral Palsy
Keywords: optic disc cupping; cerebral palsy; static encephalopathy; optic disc; optic nerve; periventricular Leukomalacia
MeSH Terms: conditions — Cerebral Palsy; Leukomalacia, Periventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Children with birth/time of neurologic insult less than 28 weeks of gestation
- 2: Children with birth/time of neurologic insult at more than 28 weeks of gestation

SUMMARY:
Hypothesis: Children born prematurely (between 8 and 9 months) with brain damage have an abnormal appearance of the optic nerve (nerve in eye) that resembles glaucoma (cupping) compared to those born before 8 months.

Purpose: to see how often children who are born prematurely and have suffered brain damage, have abnormal appearance of the optic nerve (nerve in the eye) which mimics glaucoma (cupping). This optic nerve cupping is most often seen when children are born after 8 months and is rarely seen in children born before 8 months.

Children born prematurely are known to have injuries to their brain as they are not yet fully developed. This often involves the part of the brain that involves vision. Clinicians have observed that these children have an abnormal appearance of the optic nerve (nerve in the eye), which has the appearance of glaucoma. These children often undergo extensive and often unnecessary invasive tests to rule out glaucoma. The investigators wish to establish the prevalence of this abnormality so that children are not subjected to unnecessary investigations. The investigators also want to understand how the optic nerve cupping (similar clinical picture as glaucoma) is related to the approximate timing and extent of the brain injury, the type of cerebral palsy and the motor disability of these children.

DETAILED DESCRIPTION:
This study will provide prevalence data on the occurrence of optic nerve head cupping in children with static encephalopathy in a much larger cohort than previously reported in literature (the largest cohort in literature is n=35). Children with a large optic nerve cup are treated as "glaucoma suspects". A routine glaucoma work-up in a child includes an examination under anesthesia or sedation, since children are unable to co-operate and stay still for accurate intraocular pressure measurements. These procedures often have to be periodically repeated and are a major financial burden. Importantly, they also carry substantial health risks, especially to the premature neonate who needs ICU monitoring after any anesthesia procedure. Roughly half of the children who undergo an examination under anesthesia for suspicion of glaucoma are found not to have the disease.

Children with a diagnosis of static encephalopathy attending the Pediatric Neurology clinic will be recruited. Interested patients will undergo a routine dilated eye examination after obtaining the consent and assent. The optic nerve head parameters (size, shape, color, cup-disc ratio, vessel tortuosity) will be recorded by 2 ophthalmologists experienced in the evaluation of the optic nerve. Some of the children (who are physically able to sit up in a chair and look straight ahead without blinking) will be offered disc photographs. This will be a one-time examination done during the routine clinic visit.

The prevalence of optic disc cupping (≥ 0.5) in a population of children with static encephalopathy with onset from 24-36 weeks will be obtained. Comparison of the cup/disc ratio in the 2 groups of children based on the approximate timing of the neurological insult will also be done.

The results of this study may allow pediatric ophthalmologists and glaucoma specialists to spare a child with static encephalopathy and isolated optic nerve head cupping extensive, risky and expensive glaucoma work-up.

This study will also provide more information on the patho-physiology of the developing visual nervous system.

ELIGIBILITY:
Inclusion Criteria:

* Children born prematurely at age 24-36 weeks of gestation; are currently in the age group 0-17 years and enrolled in Dr Vedanarayanan's pediatric neurology clinic.
* Diagnosis of static encephalopathy, cerebral palsy or CNS malformations
* Availability of CT head or MRI brain for review.

Exclusion Criteria:

* Parents/guardians or the child refuse consent or assent.
* Presence of ocular media opacities preventing visualization of the fundus
* The child is unable to cooperate for the ocular examination.
* Coexistent diagnosis of glaucoma
* Unable to obtain perinatal history from parents/guardians or records

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Study population will include all children attending the pediatric neurology clinic and carry a diagnosis of static encephalopathy or equivalent terms- CNS malformation syndrome or cerebral palsy.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2008-06; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Optic Disc Cupping | Initial examination

SECONDARY OUTCOMES:
Optic disc size | Inital examination

CONTACTS AND LOCATIONS:
Overall Officials: Deepta Ghate, MD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

REFERENCES:
- [Background] Jacobson L, Hellstrom A, Flodmark O. Large cups in normal-sized optic discs: a variant of optic nerve hypoplasia in children with periventricular leukomalacia. Arch Ophthalmol. 1997 Oct;115(10):1263-9. doi: 10.1001/archopht.1997.01100160433007. PMID 9338671
- [Background] Jacobson L, Hard AL, Svensson E, Flodmark O, Hellstrom A. Optic disc morphology may reveal timing of insult in children with periventricular leucomalacia and/or periventricular haemorrhage. Br J Ophthalmol. 2003 Nov;87(11):1345-9. doi: 10.1136/bjo.87.11.1345. PMID 14609830
- [Background] McLoone E, O'Keefe M, Donoghue V, McLoone S, Horgan N, Lanigan B. RetCam image analysis of optic disc morphology in premature infants and its relation to ischaemic brain injury. Br J Ophthalmol. 2006 Apr;90(4):465-71. doi: 10.1136/bjo.2005.078519. PMID 16547329
- [Background] Hellstrom A. Optic nerve morphology may reveal adverse events during prenatal and perinatal life--digital image analysis. Surv Ophthalmol. 1999 Oct;44 Suppl 1:S63-73. doi: 10.1016/s0039-6257(99)00067-3. PMID 10548118